CLINICAL TRIAL: NCT03866161
Title: The Effect of Positive Pressure Therapy (CPAP) in Patients With Obstructive Sleep Apnea on Cognitive Functions, Anxiety, and Affective Symptoms
Brief Title: The Effect of CPAP Treatment on Cognitive Functions, Anxiety, and Affective Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Milan Sova, Head of Sleep laboratory, Department of Respiratory Medicine, University Hospital Olomouc
Other Study IDs: OSAS_CPAP_CF
Record Dates: First submitted 2019-02-18; First posted 2019-03-07 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPAP group: Obstructive sleep apnea patients treated with continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure treatment

SUMMARY:
Long term, prospective study of continuous positive airway pressure treatment influence on cognitive functions in patients with obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
Brief summary:

The aim of work is to assess the extent of anxiety and affective disorders symptoms and cognitive performance in newly diagnosed patients with obstructive sleep apnea. In the second phase, follow the changes in these areas after 2 months and after 1 year of continuous treatment. The investigators can then compare the change of symptoms and cognitive performance in terms of compliance with treatment.

Course:

Recent papers discus the interconnection of anxiety and affective disorders and the deterioration of cognitive functions in patients with untreated obstructive sleep apnea. Contemporary literature also describes the effect of PAP on affective and anxiety disorders, but the results of published works are controversial and often contradictory. The effect of OSA treatment on cognitive function is explored more and studies show improvement of cognitive function while adhering to regular overpressure breathing at night. In this study patients diagnosed with OSA (Porti 7- F + G, Germany or Alice 5- Respironics, USA) indicated for PAP (AHI> 15) therapy admitted for PAP pressure adjustment will be given by investigator The Epworth Sleepiness Scale, Beck's anxiety inventory and Beck's depression inventory. Then each participant will undergo clinical examination by the investigator using Mini-International Neuropsychiatric Interview to assess whether the participant meets the ICD-10 criteria for major depressive disorder. In the next step each participant will complete three given cognitive tests (Trail making test, D2 test, Controlled Oral Word Association Test). Results of the cognitive test will be adjusted for age and compared with the population norms for each test to assess the presence of cognitive impairment at the beginning of treatment. In the next phase participants will use PAP device in the home environment for two months. At outpatient control after 2 months, participants will complete Beck's anxiety inventory and Beck's depression inventory and Epworth sleepiness scale. In the last phase participants will use PAP device for another 10 months in the home environment so the total period of treatment will be 1 year. At the outpatient control after 1 year of treatment participants will complete Beck's anxiety inventory and Beck's depression inventory and Epworth sleepiness scale, each participant will then again complete three given cognitive tests (Trail making test, D2 test, Controlled Oral Word Association Test). Information on average use over a 1-year period and compliance with treatment will be provided from the PAP device. Participants will be then divided into two groups, compliant (over 4 hours of PAP treatment per night on average) and non-compliant (less then 4 hours of PAP treatment per night on average) and the data from the questionnaires and cognitive tests will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed obstructive sleep apnea indicated for positive airway pressure therapy, i.e. Apnea-Hypopnea index AHI> 15

Exclusion Criteria:

* Psychiatric treatment
* Treatment with psychoactive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed obstructive sleep apnea indicated for positive airway pressure treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of affective symptoms after 1 year of PAP treatment | 1 year of PAP treatment
  Statistically significant change in the scores of Beck Depression Inventory.
  The total score is calculated as a sum of 21 multiple choice items. Score 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression.
Change of anxiety symptoms after 1 year of PAP treatment | 1 year of PAP treatment
  Statistically significant change in the scores of Beck Anxiety Inventory over the 1-year period of PAP treatment.
  The total score is calculated as a sum of the 21 items. Score of 0-21 = low anxiety. Score of 22-35 = moderate anxiety. Score of 36 and above = potentially concerning levels of anxiety.
Change in Controlled Oral Word Association Test after 1 year of PAP treatment | 1 year of PAP treatment
  Statistically significant change in results of Controlled Oral Word Association Test in comparison with the pre-treatment results.
  Controlled Oral Word Association Test measures spontaneous production of words beginning with some designated letter. For each of three given letters patient has 1 minute to produce as much words as possible. Total count of words will be compared, the higher count of words represents better outcome. Standardized population norms adjusted for age and education will be used to assess the results.
Change in d2 Test after 1 year of PAP treatment | 1 year of PAP treatment
  Statistically significant change in results of d2 Test in comparison with the pre-treatment results.
  d2 Test of attention is standardized test of selective and sustained attention and visual scanning speed. Results are measured as a number of mistakes made in 14 lines of symbols, in which patients mark three given symbols. Patient has 20 seconds for each line. Higher number of mistakes represents worse outcome as it points to cognitive impairment. Standardized population norms will be used to assess the results.
Change in Trail making test after 1 year of PAP treatment | 1 year of PAP treatment
  Statistically significant change in results of Trail making test in comparison with the pre-treatment results.
  Trail making test is measured in seconds as a time needed to complete trail from first to last point. Higher performing times represent worse outcomes as it points to cognitive impairment. Standardized population norms adjusted for age will be used to assess the results.

SECONDARY OUTCOMES:
Performance in Controlled Oral Word Association Test in untreated OSA patients compared to population norms. | 1 year of PAP treatment
  The results of Controlled Oral Word Association Test in OSA patients before PAP treatment will be compared with population norms to assess the cognitive impairment in untreated OSA patients.
  Controlled Oral Word Association Test measures spontaneous production of words beginning with some designated letter. For each of three given letters patient has 1 minute to produce as much words as possible. Total count of words will be compared, the higher count of words represents better outcome. Standardized population norms adjusted for age and education will be used to assess the results.
Performance in d2 Test in untreated OSA patients compared to population norms. | 1 year of PAP treatment
  The results of d2 Test in OSA patients before PAP treatment will be compared with population norms to assess the cognitive impairment in untreated OSA patients.
  d2 test of attention is standardized test of selective and sustained attention and visual scanning speed. Results are measured as a number of mistakes made in 14 lines of symbols, in which patients mark three given symbols. Patient has 20 seconds for each line. Higher number of mistakes represents worse outcome as it points to cognitive impairment. Standardized population norms will be used to assess the results.
Performance in Trail making test in untreated OSA patients compared to population norms. | 1 year of PAP treatment
  The results of Trail making test in OSA patients before PAP treatment will be compared with population norms to assess the cognitive impairment in untreated OSA patients.
  Trail making test is measured in seconds as a time needed to complete trail from first to last point. Higher performing times represent worse outcomes as it points to cognitive impairment. Standardized population norms adjusted for age will be used to assess the results.
The difference between compliant and non-compliant patients in affective symptoms after 1 year follow up. | 1 year of PAP treatment
  Statistically significant difference in the scores of Beck Depression Inventory in compliant (at least 4 hours of PAP treatment per night) and non-compliant patients (less than 4 hours of PAP treatment per night on average) after 1 year of follow up.
  The total score is calculated as a sum of 21 multiple choice items. Score 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression.
The difference between compliant and non-compliant patients in anxiety symptoms after 1 year follow up. | 1 year of PAP treatment
  Statistically significant difference in the scores of Beck Anxiety Inventory in compliant (at least 4 hours of PAP treatment per night) and non-compliant patients (less than 4 hours of PAP treatment per night on average) after 1 year of follow up.
  The total score is calculated by finding the sum of the 21 items. Score of 0-21 = low anxiety. Score of 22-35 = moderate anxiety. Score of 36 and above = potentially concerning levels of anxiety.
The difference between compliant and non-compliant patients in Controlled Oral Word Association Test after 1 year follow up. | 1 year of PAP treatment
  Statistically significant difference in the scores of Controlled Oral Word Association Test in compliant (at least 4 hours of PAP treatment per night) and non-compliant patients (less than 4 hours of PAP treatment per night on average) after 1 year of follow up.
  Controlled Oral Word Association Test measures spontaneous production of words beginning with some designated letter. For each of three given letters patient has 1 minute to produce as much words as possible. Total count of words will be compared, the higher count of words represents better outcome. Standardized population norms adjusted for age and education will be used to assess the results.
The difference between compliant and non-compliant patients in d2 Test after 1 year follow up. | 1 year of PAP treatment
  Statistically significant difference in the scores of d2 Test in compliant (at least 4 hours of PAP treatment per night) and non-compliant patients (less than 4 hours of PAP treatment per night on average) after 1 year of follow up.
  d2 test of attention is standardized test of selective and sustained attention and visual scanning speed. Results are measured as a number of mistakes made in 14 lines of symbols, in which patients mark three given symbols. Patient has 20 seconds for each line. Higher number of mistakes represents worse outcome as it points to cognitive impairment. Standardized population norms will be used to assess the results.
The difference between compliant and non-compliant patients in Trail making test after 1 year follow up. | 1 year of PAP treatment
  Statistically significant difference in the scores of Trail making test in compliant (at least 4 hours of PAP treatment per night) and non-compliant patients (less than 4 hours of PAP treatment per night on average) after 1 year of follow up.
  Trail making test is measured in seconds as a time needed to complete trail from first to last point. Higher performing times represent worse outcomes as it points to cognitive impairment. Standardized population norms adjusted for age will be used to assess the results.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Vanek, MD., Study Chair — University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bixler EO, Vgontzas AN, Lin HM, Ten Have T, Leiby BE, Vela-Bueno A, Kales A. Association of hypertension and sleep-disordered breathing. Arch Intern Med. 2000 Aug 14-28;160(15):2289-95. doi: 10.1001/archinte.160.15.2289. PMID 10927725
- [Result] Reichmuth KJ, Austin D, Skatrud JB, Young T. Association of sleep apnea and type II diabetes: a population-based study. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1590-5. doi: 10.1164/rccm.200504-637OC. Epub 2005 Sep 28. PMID 16192452
- [Result] Hobzova M, Prasko J, Vanek J, Ociskova M, Genzor S, Holubova M, Grambal A, Latalova K. Depression and obstructive sleep apnea. Neuro Endocrinol Lett. 2017 Oct;38(5):343-352. PMID 29106789
- [Result] Szaulinska K, Plywaczewski R, Sikorska O, Holka-Pokorska J, Wierzbicka A, Wichniak A, Sliwinski P. Obstructive sleep apnea in severe mental disorders. Psychiatr Pol. 2015;49(5):883-95. doi: 10.12740/PP/32566. English, Polish. PMID 26688840
- [Result] Eikermann M, Jordan AS, Chamberlin NL, Gautam S, Wellman A, Lo YL, White DP, Malhotra A. The influence of aging on pharyngeal collapsibility during sleep. Chest. 2007 Jun;131(6):1702-9. doi: 10.1378/chest.06-2653. Epub 2007 Apr 5. PMID 17413053
- [Result] Hobzova M, Hubackova L, Vanek J, Genzor S, Ociskova M, Grambal A, Prasko J. Cognitive function and depressivity before and after cpap treatment in obstructive sleep apnea patients. Neuro Endocrinol Lett. 2017 Jul;38(3):145-153. PMID 28759181
- [Derived] Vanek J, Prasko J, Genzor S, Belohradova K, Visnovsky J, Mizera J, Bocek J, Sova M, Ociskova M. Cognitive Functions, Depressive and Anxiety Symptoms After One Year of CPAP Treatment in Obstructive Sleep Apnea. Psychol Res Behav Manag. 2023 Jun 21;16:2253-2266. doi: 10.2147/PRBM.S411465. eCollection 2023. PMID 37366480